CLINICAL TRIAL: NCT00001652
Title: The Evaluation and Naturalistic Follow-up of Patients With Bipolar Disorder
Brief Title: The Evaluation and Follow-up of Patients With Bipolar Disorder
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 970039; 97-M-0039
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-12

CONDITIONS: Bipolar Disorder
Keywords: Life-Charting; Cerebrospinal Fluid; Diagnostic Tests; Cognitive Testing; Course of Illness; Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder; Disease Progression

SUMMARY:
The purpose of this research protocol is to screen and enroll individuals who have bipolar disorder and to track each person's course of illness in order to study the long-term course of illness and to elucidate possible clinical and biological predictors of acute and sustained treatment response. As a part of this protocol, subjects will: systematically be administered psychiatric rating scales such as the life-chart method (LCM) for daily assessment of mood, sleep, and behavior; be asked to participate in non-invasive research procedures, such as blood drawing for measurement of thyroid antibodies and intracellular calcium; and be medicated as is clinically appropriate. This protocol also serves as a stepping stone to other protocols such as the comparative acute and long-term efficacy of three antidepressants (#95-M-0129), and the efficacy of omega-3 fatty acids (#00-M-0004), for which separate written informed consents are obtained. Patients in this study are participants in the larger NIMH-Stanley Foundation Bipolar Network (SFBN), which involves six academic sites focused on better understanding the long-term course and treatment of the illness. The current protocol thus serves as an entry point for individuals with bipolar disorder for screening and detailed longitudinal assessment both prior to and in between more formal blind randomized IRB approved treatment protocols.

DETAILED DESCRIPTION:
The purpose of this research protocol is to screen and enroll individuals who have bipolar disorder and to track each person's course of illness in order to study the long-term course of illness and to elucidate possible clinical and biological predictors of acute and sustained treatment response. As a part of this protocol, subjects will: systematically be administered psychiatric rating scales such as the life-chart method (LCM) for daily assessment of mood, sleep, and behavior; be asked to participate in non-invasive research procedures, such as blood drawing for measurement of thyroid antibodies and intracellular calcium; and be medicated as is clinically appropriate. This protocol also serves as a stepping stone to other protocols such as the comparative acute and long-term efficacy of three antidepressants (#95-M-0129), and the efficacy of omega-3 fatty acids (#00-M-0004), for which separate written informed consents are obtained. Patients in this study are participants in the larger NIMH-Stanley Foundation Bipolar Network (SFBN), which involves six academic sites focused on better understanding the long-term course and treatment of the illness. The current protocol thus serves as an entry point for individuals with bipolar disorder for screening and detailed longitudinal assessment both prior to and in between more formal blind randomized IRB approved treatment protocols.

ELIGIBILITY:
Subjects must fulfill DSM-IV criteria for Bipolar I disorder (BPI), Bipolar II disorder (BPII), Bipolar Disorder not otherwise specified (BPNOS), or schizoaffective disorder bipolar type.

Subjects must be competent to comprehend the purpose of the study and to provide written informed consent and be willing to participate in detailed longitudinal follow-up.

Subjects will undergo complete psychiatric diagnostic interview (SCID--DSM-IV), medical, neurological, and laboratory examinations (as appropriate such as EKG, renal and liver function tests, serum electrolytes, urinalysis, HIV, hepatitis B, pregnancy testing, and urine drug screen for the presence of psychoactive drugs and drugs of abuse).

Subjects must be at least 18 years old.

Subjects should have no general medical illness that is primary (i.e. appears to be causing the mood disorder), or contraindicates the use of conventional and study medications under other protocols.

Women participants of child bearing potential must be nongravid, nonnursing, and using acceptable method of birth control such as intrauterine device, diaphragm with contraceptive foam, or condom with spermicide.

Subjects must not have alcohol or substance use or dependence of sufficient magnitude to require independent, concurrent treatment intervention (excluding self-help groups), i.e., hospitalization, day treatment programs, or counselor visits.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150
Dates: Start 1996-12; Study Completion 2002-12

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States

REFERENCES:
- [Background] Weissman MM, Leaf PJ, Tischler GL, Blazer DG, Karno M, Bruce ML, Florio LP. Affective disorders in five United States communities. Psychol Med. 1988 Feb;18(1):141-53. doi: 10.1017/s0033291700001975. PMID 3363034
- [Background] Kessler RC, McGonagle KA, Zhao S, Nelson CB, Hughes M, Eshleman S, Wittchen HU, Kendler KS. Lifetime and 12-month prevalence of DSM-III-R psychiatric disorders in the United States. Results from the National Comorbidity Survey. Arch Gen Psychiatry. 1994 Jan;51(1):8-19. doi: 10.1001/archpsyc.1994.03950010008002. PMID 8279933
- [Background] Insel TR, Kalin NH, Risch SC, Cohen RM, Murphy DL. Abducens palsy after lumbar puncture. N Engl J Med. 1980 Sep 18;303(12):703. doi: 10.1056/NEJM198009183031219. No abstract available. PMID 7402261